CLINICAL TRIAL: NCT03764540
Title: Randomized Phase II Study of Docetaxel Versus Cabazitaxel Post Abiraterone or Enzalutamide Progression
Brief Title: Docetaxel Versus Cabazitaxel Post Abiraterone or Enzalutamide
Acronym: CABPOSTAAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The cabazitaxel was recently approved by the regulatory authorities for mCRPCa
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-02-2018-7545
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; Prednisone; Docetaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cabazitaxel plus prednisone (Experimental): Cabazitaxel: Single-dose vial, containing a total of 60 mg of cabazitaxel expressed as anhydrous and solvent-free basis, per 1.5 mL of solution. Cabazitaxel will be administered by IV route Prednisone will be administered orally, 5 mg twice daily (10 mg per day total dose).
  Prednisone will be administered by oral route
  Interventions: Drug: Cabazitaxel plus prednisone
- Docetaxel plus prednisone (Active Comparator): Docetaxel is formulated in polysorbate 80 and commercially available as 80 mg/2.0 mL single-dose vials with accompanying diluent (13% ethanol in water for injection) for IV use.
  Prednisone will be administered orally, 5 mg twice daily (10 mg per day total dose).
  Prednisone will be administered by oral route
  Interventions: Drug: Docetaxel plus prednisone

INTERVENTIONS:
Drug: Cabazitaxel plus prednisone — Cabazitaxel 25 mg/m² intravenously on day 1 of each cycle, plus prednisone 10 mg orally given daily.
  A cycle is defined as a 3-weeks period for a maximum of 10 cycles.
  Other Names: Experimental
  Arms: Cabazitaxel plus prednisone
Drug: Docetaxel plus prednisone — Docetaxel 75 mg/m² intravenously on day 1 of each cycle, plus prednisone 10 mg orally given daily.
  A cycle is defined as a 3-weeks period for a maximum of 10 cycles.
  Other Names: Active Comparator
  Arms: Docetaxel plus prednisone

SUMMARY:
Prostate cancer (PCa) is the most frequently diagnosed cancer in Canadian men. While the majority of PCa is slow growing and responds well to first line treatment, a proportion of cases (10%) progress to metastatic form resulting in more than 4 000 deaths annually in Canada and 250 000 worldwide. Currently, first line treatment for PCa includes surgery, radiation and androgen deprivation therapy (ADT). A rapid evolution in the understanding of disease biology, combined with approvals of new therapies including immunotherapy, novel chemotherapy, hormonal agents and a bone calcium matrix-targeted radionuclide, along with further drugs in development, have made treatment decisions for metastatic castration-resistant prostate cancer (mCRPC) increasingly complex and challenging.

This is a Phase II Study of Cabazitaxel plus prednisone in patients with metastatic castration-resistant prostate cancer (mCRPC). The current study is designed to determine if cabazitaxel will improve progression free survival (PFS) or overall survival (OS).

This study will enroll patients with mCRPC, who have been previously treated and progressed under docetaxel or abiraterone regimen.

Patients must meet the study eligibility criteria and must be competent to give informed consent.

DETAILED DESCRIPTION:
This is a prospective, multicenter, national, randomized, open label study, comparing the efficacy of cabazitaxel at 25 mg/m² plus prednisone (Arm A) over docetaxel at 75mg/m2 plus prednisone (Arm B) after enzalutamide at 160 mg once daily or abiraterone acetate at 1000 mg once daily plus prednisone in chemotherapy-naïve patients with mCRPC who have progressed on abiraterone acetate or enzalutamide.

Each patient will be treated until disease progression, unacceptable toxicity, or patient's refusal of further study treatment.

All eligible patients will be randomly assigned to either arm A or B in a 1:1 proportion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed prostate adenocarcinoma.
* Metastatic disease.
* Progressive disease (PD) while receiving AR targeted therapy with abiraterone acetate or enzalutamide by at least one of the following:
* Progression in measurable disease (RECIST 1.1 criteria). Patient with measurable disease must have at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be at least 10 mm when measured by computed tomography (CT) [CT scan thickness no greater than 5 mm] or magnetic resonance imaging (MRI). Lymph nodes should be ≥ 15 mm in short axis. As defined by PCWG2, if lymph node metastasis is the only evidence of metastasis, it must be ≥ 20 mm in diameter when measured by spiral CT or MRI. Previously irradiated lesions, primary prostate lesion and bone lesions will be considered non-measurable disease, and/or
* Appearance of 2 or more new bone lesions. They must be confirmed by other imaging modalities (CT; MRI) if ambiguous results (PCWG2), and/or
* Rising PSA defined (PCWG2) as at least two consecutive rises in PSA to be documented over a reference value (measure 1) taken at least one week apart. The first rising PSA (measure 2) should be taken at least 7 days after the reference value. A third confirmatory PSA measure is required (2nd beyond the reference level) to be greater than the second measure and it must be obtained at least 7 days after the 2nd measure. If this is not the case, a fourth PSA measure is required to be taken and be greater than the 2nd measure. The third (or the fourth) confirmatory PSA should be taken within 4 weeks prior to randomization.
* A PSA value of at least 2 ng/mL is required at study entry.
* Effective castration (serum testosterone levels ≤0.5 ng/mL).
* Prior AR targeted therapy (abiraterone acetate or enzalutamide) must be stopped at least 2 weeks before study treatment.
* Signed written informed consent.

Exclusion Criteria:

Related to methodology:

* Prior chemotherapy for prostate cancer, except estramustine and except adjuvant/neoadjuvant treatment completed >3 years ago. Prior treatment with sipuleucel T immunotherapy is allowed at the condition patient did not received prior chemotherapy. No further anti-cancer therapy after the previous AR targeted therapy and before inclusion.
* Less than 28 days elapsed from prior treatment with radiotherapy or surgery to the time of randomization.
* Prior isotope therapy, whole bony pelvic radiotherapy, or radiotherapy to >30% of bone marrow.
* Adverse events (excluding alopecia and those listed in the specific exclusion criteria) from any prior anticancer therapy of grade >1(National Cancer Institute Common Terminology Criteria [NCI CTCAE] v4.0) at the time of randomization.
* Less than 18 years (or country's legal age of majority if the legal age is >18 years).
* Eastern Cooperative Oncology Group (ECOG) performance status >1.
* History of brain metastases, uncontrolled spinal cord compression, or carcinomatous meningitis or new evidence of brain or leptomeningeal disease.
* Prior malignancy. Adequately treated basal cell or squamous cell skin or superficial (pTis, pTa, and pT1) bladder cancer are allowed, as well as any other cancer for which treatment has been completed ≥5 years ago and from which the patient has been disease-free for ≥5 years.
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to randomization.
* Any of the following within 3 months prior to randomization: treatment resistant peptic ulcer disease, erosive esophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism, or other uncontrolled thromboembolic event.
* Acquired immunodeficiency syndrome (AIDS-related illnesses) or known HIV disease requiring antiretroviral treatment.
* Any severe acute or chronic medical condition which could impair the ability of the patient to participate to the study or interfere with interpretation of study results, or patient unable to comply with the study procedures.
* Patients with reproductive potential who do not agree to use accepted and effective method of contraception during the study treatment period and up to 6 months after the last administered dose. The definition of "effective method of contraception" will be based on the investigator's judgment.

Related to study treatment

* Known allergies, hypersensitivity or intolerance to prednisone. History of hypersensitivity to docetaxel or polysorbate 80.
* Known history of mineralocorticoid excess or deficiency.
* Unable to swallow a whole tablet or capsule
* Inadequate organ and bone marrow function as evidenced by:

  1. Hemoglobin <10.0 g/dL
  2. Absolute neutrophil count <1.5 x 109/L
  3. Platelet count <100 x 109/L
  4. AST/SGOT and/or ALT/SGPT >1.5 x ULN;
  5. Total bilirubin >1.0 x ULN
  6. Potassium <3.5 mmol/L
  7. Serum albumin <3.0 g/dL
  8. Child-Pugh Class B and C
  9. Serum Creatinine ≤ 1.5 x ULN,
* Contraindications to the use of corticosteroid treatment.
* Symptomatic peripheral neuropathy grade >2 (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v.4.0).
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 12 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or cardiac left ventricular ejection fraction (LVEF) measurement of <50% at baseline.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
PSA response rate at 6 and 12 months | through study completion, an average of 1 year
  Change from baseline PSA level of at least 50%, PSA partial response is defined as a ≥ 50% decline in PSA from cycle 1 day 1 (baseline) PSA value. This PSA change must be confirmed as sustained by a second PSA value obtained ≥ 3 weeks later.

SECONDARY OUTCOMES:
Radiological progression-free survival (rPFS) | through study completion, an average of 1 year
  Time interval between the date of randomization and the date of the first documentation of any of the following event. Radiological tumor progression by RECIST 1.1 and PCWG2,
Overall Survival | through study completion, an average of 1 year
  Time interval from the date of randomization to the date of death due to any cause
Time to PSA progression (TTPP) | through study completion, an average of 1 year
  Time interval between the date of randomization and the date of first documented PSA progression.
Tumor response | through study completion, an average of 1 year
  Measurable by RECIST 1.1
Duration of tumor response | hrough study completion, an average of 1 year
  Time between the first evaluation at which the tumor response criteria are met and the first documentation of tumor progression.
Pain response: BPI-SF pain intensity item scores | through study completion, an average of 1 year
  Decrease by <30% from baseline in the average of BPI-SF pain intensity item scores (items 3, 4, 5, and 6) observed at 2 consecutive evaluations ≥3 weeks apart without increase in analgesic usage score.
Time to Pain progression | through study completion, an average of 1 year
  Time interval between the date of randomization and the date of the first documented pain progression

CONTACTS AND LOCATIONS:
Overall Officials: fred Saad, MD, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada